CLINICAL TRIAL: NCT06682494
Title: Comparative Study on Enhancing Oral Cancer Awareness: Classical Educational Materials vs. AI-Powered Chatbot
Brief Title: Enhancing Oral Cancer Awareness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American Association for Cancer Education (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MCC-24-21890; HM20030494 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2024-10-29; First posted 2024-11-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Oral Cancer; Chatbot; Patient Education; Prevention; Oral Cancer , Oral Squamous Cell Carcinoma, Oral Cavity Cancer; Oropharyngeal Cancers
Keywords: AI-powered Chatbox; Oral cancer prevention; Socio-economic barriers
MeSH Terms: conditions — Mouth Neoplasms; Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Educational Materials (Active Comparator): Receiving oral cancer educational materials (handouts from trusted sources such as the Centers for Disease Control (CDC) and American Cancer Association (ACA) and other reliable health education resources.
  Interventions: Behavioral: Traditional Education
- Engaging with an AI-powered Chatbot (Experimental): AI-powered chatbox designed specifically for oral cancer education. The chatbot is programmed to provide accurate information on oral cancer risks, symptoms, preventive measures, and the importance of regular dental check-ups.
  Interventions: Behavioral: AI-powered Chatbox

INTERVENTIONS:
Behavioral: Traditional Education — Participants will receive traditional educational handouts focusing on increasing awareness of oral cancer risks, preventive strategies, and the importance of regular dental check-ups. Participants will be provided time to read the handouts based on calculated reading time.
  Arms: Traditional Educational Materials
Behavioral: AI-powered Chatbox — The chatbot interaction will be initiated through a provided link, allowing participants to access information and ask questions related to oral health and cancer prevention. The chatbot is programmed to provide accurate information on oral cancer risks, symptoms, preventive measures, and the importance of regular dental check-ups. Participants will be encouraged to interact with the chatbot for a specified duration
  Arms: Engaging with an AI-powered Chatbot

SUMMARY:
To evaluate the impact of AI-powered chatbot interactions versus traditional educational handouts on increasing participants' knowledge of oral cancer and its prevention

DETAILED DESCRIPTION:
The study evaluates the difference in outcome of two distinct interventions aimed at enhancing oral cancer awareness and prevention among participants from African American communities in the Richmond area. Participants assigned to the first intervention arm will receive traditional educational handouts sourced from trustworthy and reliable health sources such as the CDC, American Cancer Association (ACA), and other health education resources. These handouts will be provided to the participants and provided enough time to read them based on calculated reading time, focusing on increasing awareness of oral cancer risks, preventive strategies, and the importance of regular dental check-ups. Participants assigned to the second intervention arm will engage with an AI-powered chatbot designed specifically for oral cancer education. The chatbot interaction will be initiated through a provided link, allowing participants to access information and ask questions related to oral health and cancer prevention. The chatbot is programmed to provide accurate information on oral cancer risks, symptoms, preventive measures, and the importance of regular dental check-ups

ELIGIBILITY:
Inclusion Criteria:

* Identify as African American as defined by the US Census
* Participants must be able to read, speak, and write in English

Exclusion Criteria:

* Individuals who cannot physically or mentally participate in the research project will be excluded
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Compare participant retention rates between the AI-powered tool arm and the conventional educational material arm | Baseline, and post intervention (3 months)
  Compare the percentage of participants that continued the intervention to the participants that continued using the active comparator to measure intervention feasibility.
Evaluate the impact of AI-powered chatbot interactions versus traditional educational handouts on knowledge and behavior | Baseline, and post intervention (3 months)
  Assess the effectiveness of the interventions by baseline and post intervention surveys assessing oral cancer knowledge, attitudes, and behaviors utilizing a questionnaire based on the Health Belief Model.
  The questionnaire will include scales measuring knowledge about oral cancer, its causes, risk factors, signs, preventive methods. Each question will have one correct answer, and the final score at baseline and after the intervention will be compared. Based on previous literature, a score of 60-70% can indicate adequate knowledge about a disease, but the primary goal of the outcome is to compare improvement in knowledge between control vs intervention arms.
Investigate socio-demographic factors that affect oral cancer knowledge in the African American population | Baseline, and post intervention (3 months)
  Pre-intervention surveys will include questions assessing socio-demographic variables of the participants. These variables will serve as covariates in the analysis to measure their effects on knowledge and attitudes.
  The effect of demographic factors affecting healthcare service utilization, such as education attainment and health insurance status, on knowledge about and attitude toward oral cancer will be measured through regression analysis to investigate their impact on oral cancer awareness and prevention efforts.
Evaluate the acceptability of AI-powered chatbot interactions versus traditional educational handouts | Baseline, and post intervention (3 months)
  Assess the acceptability of the interventions by baseline and post intervention surveys assessing satisfaction, appropriateness, ease of use, and acceptability of the interventions to improve oral cancer knowledge.
  Satisfaction and acceptability will be measured through a set of questions in the post-intervention questionnaire with 5 Likert scale-based responses ranging from "Strongly Disagree" to "Strongly Agree", and the final score will be compared between arms.

CONTACTS AND LOCATIONS:
Overall Officials: Tamas Gal, Ph.D, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant survey data dictionary and individual participant responses will be shared upon request. Requests will be submitted to the PI (Tamas Gal, PhD) through email (Tamas.Gal@vcuhealth.org)
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 7/1/2025 - 6/30/2030
Access Criteria: Data will be shared upon request. Requests will be submitted to the PI (Tamas Gal, PhD) through email (Tamas.Gal@vcuhealth.org)